CLINICAL TRIAL: NCT04647916
Title: A Phase II Trial of Sacituzumab Govitecan (IMMU-132) (NSC #820016) for Patients With HER2-Negative Breast Cancer and Brain Metastases
Brief Title: Testing Sacituzumab Govitecan Therapy in Patients With HER2-Negative Breast Cancer and Brain Metastases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S2007; NCI-2020-07706 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); S2007 (Other: SWOG); S2007 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Invasive Breast Carcinoma; Metastatic HER2 Negative Breast Carcinoma; Metastatic Malignant Neoplasm in the Brain; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Brain Neoplasms | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (sacituzumab govitecan) (Experimental): Patients receive sacituzumab govitecan IV over 1-3 hours on days 1 and 8. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Sacituzumab Govitecan

INTERVENTIONS:
Biological: Sacituzumab Govitecan — Given IV
  Other Names: hRS7-SN38 Antibody Drug Conjugate; IMMU-132; RS7-SN38; Sacituzumab Govitecan-hziy; Trodelvy

SUMMARY:
This phase II trial studies the effect of sacituzumab govitecan in treating patients with HER2-negative breast cancer that has spread to the brain (brain metastases). Sacituzumab govitecan is a monoclonal antibody, called sacituzumab, linked to a chemotherapy drug, called govitecan. Sacituzumab is a form of targeted therapy because it attaches to specific molecules on the surface of cancer cells, known as Trop-2 receptors, and delivers govitecan to kill them. Giving sacituzumab govitecan may shrink the cancer in the brain and/or extend the time until the cancer gets worse.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the intracranial objective response rate (ORR) (complete response [CR] or partial response [PR] by Response Assessment in Neuro-Oncology Brain Metastases [RANO-BM]) with sacituzumab govitecan (IMMU-132) in patients with HER2-negative metastatic breast cancer with brain involvement.

SECONDARY OBJECTIVES:

I. To evaluate bi-compartmental progression-free survival in this population. II. To evaluate overall survival in this population. III. To assess safety and tolerability of sacituzumab govitecan (IMMU-132) treatment in this population.

IV. To evaluate ORR by hormone-receptor (HR) subgroup (HR+, HR-).

BANKING OBJECTIVE:

I. To bank specimens for future correlative studies.

OUTLINE:

Patients receive sacituzumab govitecan intravenously (IV) over 1-3 hours on days 1 and 8. Cycles repeat every 21 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study registration, patients are followed up every 3 months for 1 year and then every 6 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed HER2-negative (per 2018 American Society of Clinical Oncology [ASCO]/College of American Pathologists [CAP] joint guideline) invasive breast cancer that has metastasized to the brain. NOTE: Pathology report must confirm HER2-negative invasive breast cancer. Brain metastases must be confirmed by radiology report
* Participants must have an magnetic resonance imaging (MRI) of the brain within 28 days prior to registration and must have central nervous system metastases with at least one measurable brain metastasis >= 1.0 cm in size (per RANO-BM) that has not been irradiated, or has progressed despite prior radiation therapy (in the opinion of the treating physician). In the rare case that a previously irradiated brain metastasis is the sole target lesion and if there is concern about possible radiation necrosis, patient is eligible only if there is clear progression in the previously radiated lesion. Computed tomography (CT) of the head cannot substitute for brain MRI. All central nervous system (CNS) disease must be assessed and documented on the S2007 Brain Metastases Baseline Tumor Assessment Form
* Participants may have measurable or non-measurable extracranial disease. All measurable disease must be assessed within 28 days prior to registration; all non-measurable disease must be assessed within 42 days prior to registration. Participants are NOT required to have extracranial disease, but must have scans done to document disease status at baseline. All extracranial disease must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1). NOTE: Brain lesions should not be included on the Baseline Tumor Assessment Form (RECIST 1.1) for this study
* Participants must have had CNS progression after previous CNS-directed therapy (radiation therapy, surgery, or any combination of therapy)
* Participants must have resolution of adverse event(s) of the most recent prior systemic anti-cancer therapy to < grade 2, with the exception of alopecia and =< grade 2 neuropathy, which are allowed
* Participants with a prior or concurrent malignancy whose natural history or treatment (in the opinion of the treating physician) does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Participants must have Zubrod performance status 0 or 1
* Participants must have history and physical exam obtained within 21 days prior to registration
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained within 21 days prior to registration)
* Platelet count >= 100,000/mcL (obtained within 21 days prior to registration)
* Hemoglobin >= 9.0 g/dL (obtained within 21 days prior to registration)
* Total bilirubin =< 1.5 times institutional upper limit of normal (ULN) (obtained within 21 days prior to registration)
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x institutional ULN (obtained within 21 days prior to registration)
* Participants must have a serum creatinine =< 1.5 times the institutional upper limit of normal (IULN) OR measured OR calculated creatinine clearance >= 30 mL/min using the following Cockcroft-Gault Formula. This specimen must have been drawn and processed within 21 days prior to registration
* Participants must have adequate cardiac function. Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, must have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification, and must be class 2B or better
* Participants must be offered the opportunity to participate in specimen banking. With participant consent, specimens must be collected and submitted via the Southwest Oncology Group (SWOG) Specimen Tracking System
* Participants must be informed of the investigational nature of this study and must sign and give informed consent in accordance with institutional and federal guidelines

Exclusion Criteria:

* Participants must not have had more than 2 seizures within 28 days prior to registration
* Participants must not have received systemic therapy (including small-molecule kinase inhibitors) or non-cytotoxic hormonal therapy (e.g., tamoxifen) within 7 days prior to registration
* Participants must not have received anti-cancer biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to registration
* Participants must not have received nitrosoureas or mitomycin C within 42 days, metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days prior to registration
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral agents that are strong CYP3A4 inhibitors or inducers and who are unwilling or unable to change to antiretroviral therapies without such interactions are ineligible because of the potential for pharmacokinetic interactions with sacituzumab govitecan (IMMU-132)
* Due to potential drug interactions of anti-retroviral drugs with sacituzumab govitecan (IMMU-132), participants must not have known active or chronic hepatitis B virus (HBV) infection, requiring suppressive therapy or known active hepatitis C virus (HCV) infection. Participants with a known history of HCV infection must have been treated and cured
* Participants must not have received enzyme-inducing anti-epileptic agents (e.g., carbamazepine, phenytoin, phenobarbital, primidone) within 7 days prior to registration or within 14 days of planned start of cycle 1, day 1 treatment, and participants must not be planning to receive enzyme-inducing anti-epileptic agents (e.g., carbamazepine, phenytoin, phenobarbital, primidone) for the duration of protocol treatment
* Participants must not be receiving warfarin (or other coumarin derivatives) at time of registration or be planning to receive warfarin (or other coumarin derivatives) for the duration of protocol treatment. Participants who are able to switch to low molecular weight heparin (LMWH) or direct oral anticoagulants (DOACs) prior to date of registration (and plan to remain off of warfarin or other coumarin derivatives) for the duration of protocol treatment) are eligible
* Patients must not be receiving or be planning to receive concomitantly any other anti-cancer therapy, including endocrine therapy. Note: Concomitant hormone replacement therapy is allowed
* Participants must not have a condition requiring ongoing systemic treatment with corticosteroids (> 4 mg daily dexamethasone [or bioequivalent]) or other immunosuppressive medications within 7 days prior to the baseline MRI. Corticosteroids administration must be stable and planned to remain =< 4 mg daily for the duration of protocol treatment. However, use of corticosteroids for clinical symptoms is allowed based upon treating physician discretion
* Participants must not have uncontrolled diabetes in the opinion of the treating investigator 21 days prior to registration
* Participants must not be pregnant or nursing. Women of reproductive potential must have a negative serum or urine pregnancy test within 7 days prior to registration. Women and men of reproductive potential must have agreed to use an effective contraceptive method for the duration of protocol treatment and for at least 6 months after the last dose of sacituzumab govitecan (IMMU-132). A woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months. In addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation. However, if at any point a previously celibate participant chooses to become heterosexually active during the time period for use of contraceptive measures outlined, he/she is responsible for beginning contraceptive measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2021-06-08 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  ORR will be evaluated using use a Simon two-stage minimax design.

SECONDARY OUTCOMES:
Overall survival | From date of registration to date of death due to any cause, assessed up to 2 years
  Will use the Kaplan-Meier curves to estimate the respective survival curves.
Progression-free survival | From date of registration to date of first documentation of progression or symptomatic deterioration or death due to any cause, assessed up to 2 years
  Will use the Kaplan-Meier curves to estimate the respective survival curves.
Incidence of adverse events | Up to 2 years
  Adverse events will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. The incidence of adverse events will be reported. Toxicity will be by grade and attribution to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Brenner, Principal Investigator — SWOG Cancer Research Network
Locations (296):
- United States (296):
  - Anchorage Associates in Radiation Medicine, Anchorage, Alaska
  - Anchorage Radiation Therapy Center, Anchorage, Alaska
  - Alaska Breast Care and Surgery LLC, Anchorage, Alaska
  - Alaska Oncology and Hematology LLC, Anchorage, Alaska
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Anchorage Oncology Centre, Anchorage, Alaska
  - Katmai Oncology Group, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - University of Arizona Cancer Center-Orange Grove Campus, Tucson, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - UC Irvine Health Cancer Center-Newport, Costa Mesa, California
  - Epic Care-Dublin, Dublin, California
  - Bay Area Breast Surgeons Inc, Emeryville, California
  - Epic Care Partners in Cancer Care, Emeryville, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Tumor Institute, Oakland, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Saint John's Cancer Institute, Santa Monica, California
  - Epic Care Cyberknife Center, Walnut Creek, California
  - Rocky Mountain Cancer Centers-Aurora, Aurora, Colorado
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Foothills Hospital, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers - Centennial, Centennial, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - The Women's Imaging Center, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Cancer Centers-Midtown, Denver, Colorado
  - Rocky Mountain Cancer Centers-Rose, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Western Surgical Care, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center - Swedish, Englewood, Colorado
  - Rocky Mountain Cancer Centers - Swedish, Englewood, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - The Melanoma and Skin Cancer Institute, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Rocky Mountain Cancer Centers-Littleton, Littleton, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Rocky Mountain Cancer Centers-Sky Ridge, Lone Tree, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Illinois CancerCare-Dixon, Dixon, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC - Ames, Ames, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Saint Anthony Regional Hospital, Carroll, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - Trinity Regional Medical Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Central Care Cancer Center - Garden City, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - HaysMed University of Kansas Health System, Hays, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Olathe Health Cancer Center, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Ascension Via Christi - Pittsburg, Pittsburg, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Hickman Cancer Center, Adrian, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Toledo Clinic Cancer Centers-Monroe, Monroe, Michigan
  - Ascension Providence Hospitals - Novi, Novi, Michigan
  - Ascension Providence Hospitals - Southfield, Southfield, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Golden Triangle, Columbus, Mississippi
  - Baptist Cancer Center-Grenada, Grenada, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Saint Louis Cancer and Breast Institute-Ballwin, Ballwin, Missouri
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Capital Region Southwest Campus, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Centers, Kansas City, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Solinsky Center for Cancer Care, Manchester, New Hampshire
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - Good Samaritan Hospital Medical Center, West Islip, New York
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physician LLC-Miami Valley Hospital North, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - South Pointe Hospital, Warrensville Heights, Ohio
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Saint Charles Health System, Bend, Oregon
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Bay Area Hospital, Coos Bay, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Saint Charles Health System-Redmond, Redmond, Oregon
  - UPMC Camp Hill, Camp Hill, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - UPMC-Mercy Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - MGC Hematology Oncology-Union, Union, South Carolina
  - Baptist Memorial Hospital and Cancer Center-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Providence Regional Cancer System-Aberdeen, Aberdeen, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Providence Regional Cancer System-Centralia, Centralia, Washington
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Providence Regional Cancer Partnership, Everett, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Swedish Cancer Institute-Issaquah, Issaquah, Washington
  - Kadlec Clinic Hematology and Oncology, Kennewick, Washington
  - Providence Regional Cancer System-Lacey, Lacey, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - PeaceHealth Saint John Medical Center, Longview, Washington
  - Jefferson Healthcare, Port Townsend, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Pacific Gynecology Specialists, Seattle, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Swedish Medical Center-Cherry Hill, Seattle, Washington
  - PeaceHealth United General Medical Center, Sedro-Woolley, Washington
  - Providence Regional Cancer System-Shelton, Shelton, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Providence Regional Cancer System-Yelm, Yelm, Washington
  - Cheyenne Regional Medical Center-West, Cheyenne, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Kwapisz D. Sacituzumab Govitecan-hziy in Breast Cancer. Am J Clin Oncol. 2022 Jul 1;45(7):279-285. doi: 10.1097/COC.0000000000000919. Epub 2022 May 12. PMID 35728046